CLINICAL TRIAL: NCT01757405
Title: A PHASE 3, PROSPECTIVE, OPEN-LABEL, RANDOMIZED STUDY TO EVALUATE SAFETY AND EFFICACY OF RECOMBINANT ACTIVATED FVII BI (rFVIIa BI) IN THE TREATMENT OF ACUTE BLEEDING EPISODES PER AN ON-DEMAND REGIMEN IN PATIENTS WITH HEMOPHILIA A OR B WITH INHIBITORS
Brief Title: Recombinant Factor VIIa BI (rFVIIa BI) Treatment of Acute Bleeding Episodes Per an On-demand Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 021101; 2011-006294-26 (EudraCT Number)
Record Dates: First submitted 2012-12-21; First posted 2012-12-28 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: with Factor VIII (FVIII) or Factor IX (FIX) inhibitors
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ≤ 3 doses of 90 µg/kg rFVIIa BI (Experimental)
  Interventions: Biological: Recombinant Factor VIIa BI (rFVIIa BI)
- One dose of 270 µg/kg rFVIIa BI (Experimental)
  Interventions: Biological: Recombinant Factor VIIa BI (rFVIIa BI)

INTERVENTIONS:
Biological: Recombinant Factor VIIa BI (rFVIIa BI) — Administered approximately every 3 hours as an intravenous bolus injection on-demand
  Arms: ≤ 3 doses of 90 µg/kg rFVIIa BI
Biological: Recombinant Factor VIIa BI (rFVIIa BI) — Administered as a single intravenous bolus injection on-demand
  Arms: One dose of 270 µg/kg rFVIIa BI

SUMMARY:
The purpose of the study is to determine the efficacy and safety of rFVIIa BI as part of a six-month on-demand treatment regimen in hemophilia A or B subjects with inhibitors.

ELIGIBILITY:
Main Inclusion Criteria:

* Participant is male with hemophilia A or B with inhibitors, with a high titer (≥5 Bethesda unit (BU)) or a historical high anamnestic response.
* Participant is 12 to 65 years old at the time of screening.
* Participant is currently using or has used bypassing agents for treatment of bleeding episodes.
* Participant has an annualized bleed rate of 5 or more bleeding episodes per year on average over the 2 years prior to the Screening visit.
* Participant has a Karnofsky Performance Score ≥60.
* Participant is hepatitis C virus negative (HCV-) either by antibody testing or polymerase chain reaction (PCR); or hepatitis C virus positive (HCV+) with stable hepatic disease.
* Participant is human immunodeficiency virus negative (HIV-) or HIV+ with stable disease, CD4+ count ≥200 cells/mm^3 at screening.
* Participant is willing and able to comply with the requirements of the protocol.

Main Exclusion Criteria:

* Participant is not willing to go on an on-demand treatment scheme.
* Participant is positive for a FVII inhibitor at screening.
* Participant has clinically symptomatic liver disease.
* Participant has a platelet count <100,000/µL.
* The use of α-interferon with or without ribavirin is planned for an HCV-infected participant or the use of a protease inhibitor is planned for an HIV-infected participant.

  * Participants currently taking any of these medications for ≥30 days are eligible.
* Participant has a known hypersensitivity to rFVIIa, hamster or murine proteins, or Tween 80.
* Participant has a known history of being non-responsive to rFVIIa treatment of bleeding episodes.
* Participant has a prior history of thromboembolic event or diagnosis of other diseases that may increase the participant's risk of thromboembolic complications.
* Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
* Participant is a family member or employee of the investigator.
* Participant is scheduled for surgery during the study period.

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2014-11-11 (Actual); Study Completion 2014-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (16):
- Health Point Medical Group "St Joseph's Children's Hospital", Tampa, Florida, United States
- Japan (2):
  - Nara Medical University Hospital, Nara
  - Tokyo Medical University Hospital, Tokyo
- Poland (2):
  - Kracow Medical Center, LLC, Krakow
  - Institute of Haematology and Transfusion Medicine, Clinic of Haemostatic Disorders and Internal Diseases, Warsaw
- Louis Turcanu Emergency Clinical Children´s Hospital, Timișoara, Romania
- Russia (3):
  - Kirov Hematology and Blood Transfusion Research Institute under the Federal Medical and Biological Agency of Russia, Kirov
  - Hematology Research Center under RAMS (State Institution), Department of Reconstructive Orthopedic Surgery for Hemophilia Patients, Moscow
  - St. Petersburg City Healthcare Institution Municipal Policlinic # 37, Saint Petersburg
- Clinic for Hematology of the Clinical Center of Serbia, Belgrade, Serbia
- Spain (2):
  - Hospital Teresa Herrera Materno Infantil del C.H.U.Carretera del Pasajes/nlaboratorio de hematología, A Coruña
  - University Hospital Virgen del Rocio, Seville
- Tri-Service General Hospital (TSGH), Taipei, Taiwan
- Ukraine (3):
  - V.K. Gusak Institute of Urgent and Reconstructive Surgery within the Ukrainian National Academy of Medical Sciences, Hematology Department, Donetsk
  - Kyiv City Clinical Hospital #9, City Scientific-Practical Center for Diagnostics and Treatment of Patients with Hemostatic Pathlogies, Kiev
  - State Institution "Institute of Blood Pathology and Transfusion Medicine within the Ukrainian National Academy of Medical Sciences", Hematology Department, Lviv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conduced at 16 clinical sites from the following countries: Japan, Taiwan, Poland, Romania, Russian Federation, Serbia, Spain, Ukraine and the United States.
Pre-assignment Details: 40 participants provided informed consent and were screened for study participation, of which there was 1 screen failure. 39 participants (in pre-assignment period) were randomized where 1 participant withdrew after randomization but prior to treatment, therefore 38 participants were treated with recombinant activated factor VII BI (rFVIIa).
Groups:
- Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI: Bleeding episodes treated with up to 3 doses of 90 micrograms/kg of recombinant activated factor VII BI (rFVIIaBI) every 3 hours as on-demand intravenous bolus infusions.
- Arm 2: 1 x 270 Micrograms/kg rFVIIa BI: Bleeding episodes treated with 1 dose of 270 micrograms/kg of recombinant activated factor VII BI (rFVIIa BI) as on-demand intravenous bolus infusion.
Period: Overall Study
Arm/Group | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI
Started | 18 | 20
Completed | 17 | 18
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Median (Full Range); unit: Years] | 28 [12 to 53] | 28 [12 to 54] | 28 [12 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Bleeding Episode With "Treatment Success"
Description: No additional hemostatic product required within 12 hours of first dose other than the prescribed dosing regimen.
Time Frame: within 12 hours of first dose
Population: Full Analysis Dataset
Measure: Number (95% Confidence Interval); unit: percent of bleeding episodes
Units Other Than Participants: Bleeding Episodes
Arm/Group | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI
Number analyzed (Participants) | 18 | 20
Number analyzed (Bleeding Episodes) | 289 | 256
percent of bleeding episodes | 96.19 [93.31 to 97.86] | 79.30 [73.92 to 83.81]
Statistical Analysis 1: Comparison: Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI vs Arm 2: 1 x 270 Micrograms/kg rFVIIa BI; Equivalence test of successfully treated bleeding episodes (BEs) between or within treatment arms. Denoting the success rates in the two treatment groups by p1 and p2 , the null hypotheses of H01 : p1/p2 < 0.83 and H02 : p1/p2 > 1.20 was implicitly tested against the one-sided alternatives Ha1: 0.83 ≤ p1/p2 and Ha2 : p1/p2 ≤ 1.20, by comparing the 90% two-sided confidence interval (CI) of the ratio of success proportions to the equivalence region defined as [0.83, 1.20]; Test type: Non-Inferiority or Equivalence — Equivalence of treatment success proportions in all bleeding episodes for the two treatment groups was determined by comparing the 90% two-sided CI of the ratio of success proportions to the equivalence region defined as [0.83, 1.20]; Ratio of success proportion; Ratio of success proportion = 1.21, 90% CI 2-sided [1.15 to 1.28]

2. Secondary Outcome: Treatment Response for Each Bleeding Episode
Description: Participants rated the treatment of each bleeding episode. If treatment occurred under direct supervision of treating physician, the physician rated the response. Ratings based on a 4 point scale; EXCELLENT - full relief of pain and cessation of objective signs of bleeding (swelling, tenderness, decrease in range of motion [for muscle bleeds]) within 9 hours of treatment initiation. No additional infusion required to control bleeding, other than prescribed dosing regimen. GOOD - Substantial relief of pain and/or cessation of objective signs of bleeding within 9 hours of treatment initiation. No additional infusion required to control bleeding, other than prescribed dosing regimen. MODERATE - slight relief of pain and slight improvement of signs of bleeding within 9 hours of treatment initiation. Requires additional infusion beyond treatment regimen. NONE - No improvement or condition worsens. SUCCESSFUL = EXCELLENT or GOOD.
Time Frame: within 24 hours of infusion
Population: Full Analysis Dataset
Measure: Number (95% Confidence Interval); unit: percent of bleeding episodes
Units Other Than Participants: Bleeding Episodes
Arm/Group | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI
Number analyzed (Participants) | 18 | 20
Number analyzed (Bleeding Episodes) | 289 | 256
percent of bleeding episodes
  Successful | 87.89 [83.62 to 91.16] | 79.30 [73.92 to 83.81]
  Excellent | 34.60 [29.35 to 40.26] | 36.72 [31.05 to 42.78]
  Good | 53.29 [47.53 to 58.96] | 42.58 [36.67 to 48.70]
  Moderate | 9.69 [6.79 to 13.65] | 18.36 [14.10 to 23.56]
  No Assessment Available | 0 [0 to 0] | 0.39 [0.07 to 2.18]
  None | 2.42 [1.18 to 4.91] | 1.95 [0.84 to 4.49]

3. Secondary Outcome: Percentage of Clinical Responders (Sustained Bleeding Control) for All Acute Bleeding Episodes
Description: Clinical responders defined as sustained bleeding control, (no additional hemostatic medication including rFVIIa BI required between 12 and 24 hours after first infusion of the successfully treated bleeding episode).
Time Frame: 24 hours post infusion
Population: Full Analysis Dataset
Measure: Number (95% Confidence Interval); unit: percent of bleeding episodes
Units Other Than Participants: Bleeding Episodes
Arm/Group | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI
Number analyzed (Participants) | 18 | 20
Number analyzed (Bleeding Episodes) | 289 | 256
percent of bleeding episodes | 93.43 [89.96 to 95.75] | 76.17 [70.59 to 80.98]

4. Secondary Outcome: Safety and Tolerability of Treatment Regimens by Clinical Assessment of Percentage of Participants With Adverse Events (AEs)
Description: Safety was determined by the number of AEs (both serious AEs [SAEs] and non-serious AEs [nsAE]). Tolerability was determined by the number of AEs related to rFVIIa BI (both SAEs and nsAEs) as determined by causality assessment of the AEs by the investigator. An AE was deemed Related if the investigator judged the AE to be "possibly related" or "probably related" to rFVIIa BI. The percentage of participants with AEs were presented by seriousness (SAE, nsAE), severity (Mild, Moderate or Severe) and causality (Related or Not Related to rFVIIa BI).
Time Frame: 6 months (throughout study period)
Population: Safety Analysis Dataset
Measure: Number; unit: percent of participants with AEs
Arm/Group | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI
Number analyzed (Participants) | 18 | 20
percent of participants with AEs
  SAE-Moderate-Unrelated | 5.6 | 5.0
  SAE-Severe-Unrelated | 11.1 | 0
  SAE-Severe-Related | 0 | 5.0
  nsAE-Mild-Unrelated | 22.2 | 30.0
  nsAE-Moderate-Unrelated | 0 | 15.0

5. Secondary Outcome: Safety and Tolerability of Treatment Regimens by Clinical Assessment of Adverse Events (AEs)
Description: Safety was determined by the number of AEs (both serious AEs [SAEs] and non-serious AEs [nsAE]). Tolerability was determined by the number of AEs related to rFVIIa BI (both SAEs and nsAEs) as determined by causality assessment of the AEs by the investigator. An AE was deemed Related if the investigator judges the AE to be "possibly related" or "probably related" to rFVIIa BI. The percentage of AEs were presented by seriousness (SAE, nsAE), severity (Mild, Moderate or Severe) and causality (Related or Not Related [to rFVIIa BI]).
Time Frame: 6 months (throughout study period)
Population: Safety Analysis Dataset
Measure: Number; unit: percent of AEs
Units Other Than Participants: adverse events
Arm/Group | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI
Number analyzed (Participants) | 18 | 20
Number analyzed (adverse events) | 15 | 16
percent of AEs
  SAE-Moderate-Unrelated | 6.7 | 6.3
  SAE-Severe-Unrelated | 20.0 | 0
  SAE-Severe-Related | 0 | 12.5
  nsAE-Mild-Unrelated | 73.3 | 62.5
  nsAE-Moderate-Unrelated | 0 | 18.8

6. Secondary Outcome: Percentage of Participants With Inhibitor Development to FVII
Description: Development of rFVII inhibitors or FVIIa binding antibodies during the study.
Time Frame: 6 months (throughout study period)
Population: Safety Analysis Dataset
Measure: Number; unit: percent of participants
Arm/Group | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI
Number analyzed (Participants) | 18 | 20
percent of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months (throughout study period)
Groups:
- Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI: Bleeding episodes treated with up to 3 doses of 90 micrograms/kg of recombinant activated factor VII BI (rFVIIa BI) every 3 hours as on-demand intravenous bolus infusions.
Arm/Group | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI
Serious Adverse Events (participants affected / at risk) | 2/18 | 2/20
Other Adverse Events (participants affected / at risk) | 4/18 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI (N=18) | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI (N=20)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug Ineffective (General disorders) | 0 (0) | 1 (1)
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: up to 3 x 90 Micrograms/kg rFVIIa BI (N=18) | Arm 2: 1 x 270 Micrograms/kg rFVIIa BI (N=20)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Sinus Headache (Nervous system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Tinea Versicolour (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, results may not be published without prior written approval of Sponsor.